CLINICAL TRIAL: NCT04797260
Title: Phase I/II Clinical Trial of Autologous Hematopoietic Stem Cell Gene Therapy in RAG1-Deficient Severe Combined Immunodeficiency
Brief Title: Phase I/II Clinical Trial Stem Cell Gene Therapy in RAG1-Deficient SCID
Acronym: RAG1-SCID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Horizon 2020 - European Commission (Other)
Responsible Party: Principal Investigator, alankester, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L20.067
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Severe Combined Immunodeficiency Due to RAG1 Deficiency
Keywords: SCID; RAG1; Gene Therapy
MeSH Terms: interventions — Genetic Therapy

STUDY DESIGN:
Intervention Model Description: CD34+ HSC from patient will be obtained by leukapheresis or from bone marrow. After purification, CD34+ cells will be transduced with the SIN-LV-RAG1 vector. Transduced cells will be cryopreserved. Upon confirmation of successful transduction and meeting the release criteria as RAG1 LV CD34+ cells, patient conditioning will be allowed to start. After patient conditioning, cryopreserved RAG1 LV CD34+ cells will be thawed and administered to the patient. In case of failure of hematopoietic reconstitution after infusion of the RAG1 LV CD34+ cells the autologous backup graft will be infused to rescue the patient from aplasia. In addition, a conventional allogeneic HSCT procedure will be scheduled. Patients included in this study will be monitored on protocol during the first two years after infusion of the RAG1 LV CD34+ cells as per study protocol. Follow up as part of the routine clinical care for post-transplant patients will be annual after this, for at least 15 years after infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gene therapy (Experimental): In this arm, 10 patients will be included for gene therarpy
  Interventions: Genetic: Gene therapy

INTERVENTIONS:
Genetic: Gene therapy — Patients will be infused with autologous CD34+ cells transduced with the pCCL.MND.coRAG1.wpre lentiviral vector (RAG1 LV CD34+ cells).

SUMMARY:
This study is a prospective, non-randomized, open-label, two-centre phase I/II intervention study designed to treat children up to 24 months of age with RAG1-deficient SCID with an indication for allogeneic hematopoietic stem cell transplantation but lacking an HLA-matched donor. The study involves infusion of autologous CD34+ cells transduced with the pCCL.MND.coRAG1.wpre lentiviral vector (hereafter called RAG1 LV CD34+ cells) in five patients with RAG1-deficient SCID.

DETAILED DESCRIPTION:
Severe combined immunodeficiency (SCID) is a genetically heterogeneous life-threatening disease characterized by severely impaired T cell development with or without impaired natural killer (NK) and B cell development or function depending on the genetic defect. Mutations in recombination activating genes 1 and 2 (RAG1 and RAG2) represent about 20% of all types of SCID. SCID is a paediatric emergency since it leads to severe and recurrent infections often in combination with protracted diarrhoea and failure to thrive. When left untreated, it is usually fatal within the first year of life. Currently, the only curative treatment option for RAG-deficient SCID is allogeneic hematopoietic stem cell transplantation (HSCT). Despite improvements in HSCT in recent years, this treatment is associated with serious potential complications like graft-versus-host disease which results in an unfavourable outcome, particularly in patients who lack a human leukocyte antigen (HLA)-matched donor. In recent years, gene therapy based on transplantation of autologous gene-corrected hematopoietic stem cells (HSC) has evolved as an effective and safe therapeutic option for X-linked and ADA-deficient forms of SCID. We have recently demonstrated that gene therapy using lentiviral (LV) self-inactivating (SIN) vectors expressing codon-optimized human RAG1 in a mouse model for RAG1-deficient SCID effectively restores T and B cell development and function. In this phase I/II explorative intervention study feasibility, safety and efficacy of gene therapy using gene-corrected autologous CD34+-selected mobilized peripheral blood or bone marrow cells will be investigated in patients with RAG1-deficient SCID with an indication for allogeneic HSCT but lacking an human leukocyte antigen (HLA)-matched donor.

ELIGIBILITY:
Inclusion Criteria:

1. RAG1-deficient SCID as confirmed by genetic analysis
2. Peripheral blood T cells < 300/μL and/or naïve T cells < 1/μL
3. Age < 2 years
4. Age at least 8 weeks by the time of busulfan and fludarabine administration
5. Lack of an available HLA-matched donor (HLA-identical sibling or 10/10 (A, B, C, DR, DQ) allele-matched (un)related donor)
6. Signed informed consent (parental or guardian)
7. Able to return to the study centre for follow-up (per protocol) during the 2-year study and the 15-year long-term off study review

Exclusion Criteria:

1. Availability of an HLA-matched donor (HLA-identical sibling or 10/10 (A, B, C, DR, DQ) allele-matched (un)related donor)
2. RAG1 deficiency with peripheral blood T cells > 300/μL and/or naïve T cells > 1/μL
3. Omenn syndrome
4. Previous allogeneic HSCT
5. Significant organ dysfunction/co-morbidity (including but not limited to the ones listed below):

   1. Mechanical ventilation
   2. Shortening fraction on echocardiogram <25%
   3. Renal failure defined as dialysis dependence
   4. Uncontrolled seizure disorder
6. Any other condition that the investigator considers is a contraindication to collection and/or infusion of trans-duced cells for that individual or indicate patient's inability to follow the protocol, for example contraindication f to busulfan, major congenital abnormalities, ineligible to receive anaesthesia, or documented refusal or inability of the family to return for scheduled visits.
7. Human immunodeficiency virus (HIV) infection or Human T-cell Leukemia Virus (HTLV) infection

Ages: 8 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of successful generation of RAG1 LV CD34+ cells | 2 years
  IMP (RAG1 LV CD34+ cells) that meets the release criteria as defined in the IMPD.
Safety of RAG1 lentiviral gene therapy | 2 years
  Overall survival and event-free survival (EFS) after infusion of the IMP with events

SECONDARY OUTCOMES:
T cell reconstitution | 1 year
  CD3 T cells > 300/μL and CD4 > 200/μL at 1 year
Thymic function | 1 year
  presence of naïve CD4 T cells at 1 year
T and B cell receptor repertoire | 1 year
  Molecular T and B cell receptor repertoire at 1 year
Immunoglobulin dependence | 2 years
  Immunoglobulin supplementation dependence at 2 years
Persistence of gene marking | 1 year
  Gene marking in myeloid and lymphoid lineages in blood at six months and one year and in bone marrow at one year
Occurrence of Infections | 2 years
  Frequency of serious/invasive infections
Failure to thrive | 2 years
  Recovery from failure to thrive
Quality of life | 2 years
  Quality of life at 2 years (assessed using PedsQL by proxy).

CONTACTS AND LOCATIONS:
Overall Officials: Arjan C Lankester, Prof.dr., Principal Investigator — Leiden University Medical Center
Locations (7):
- The Royal Childrens Hospital, Melbourne, Australia
- Ospedale Pediatrico Bambino Gesù, Roma, Italy
- Leiden University Medical Center, Leiden, Netherlands
- Wroclaw Medical University, Wroclaw, Poland
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Erciyes Üniversitesi TIP Fakültesi, Kayseri, Turkey (Türkiye)
- University College London Great Ormond Street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia-Perez L, van Eggermond M, van Roon L, Vloemans SA, Cordes M, Schambach A, Rothe M, Berghuis D, Lagresle-Peyrou C, Cavazzana M, Zhang F, Thrasher AJ, Salvatori D, Meij P, Villa A, Van Dongen JJM, Zwaginga JJ, van der Burg M, Gaspar HB, Lankester A, Staal FJT, Pike-Overzet K. Successful Preclinical Development of Gene Therapy for Recombinase-Activating Gene-1-Deficient SCID. Mol Ther Methods Clin Dev. 2020 Mar 31;17:666-682. doi: 10.1016/j.omtm.2020.03.016. eCollection 2020 Jun 12. PMID 32322605